CLINICAL TRIAL: NCT02724540
Title: Randomized Embolization Trial for NeuroEndocrine Tumor Metastases to the Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 01215
Record Dates: First submitted 2016-03-28; First posted 2016-03-31 (Estimated); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Neuroendocrine Tumor, Malignant; Liver Metastases
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (3):
- Arm 1 - BE (Experimental): Lobar or segmental bland embolization (BE) with microspheres (50-500 microns) to 2-5 heartbeat stasis.
  Interventions: Device: Bland Embolization
- Arm 2 - TACE (Experimental): Lobar or segmental lipiodol conventional transarterial chemoembolization (TACE). Doxorubicin 50 mg dissolved in 10 mL dilute contrast and emulsified with 10-20 cc iodized oil, followed by 50-500 μm microspheres.
  Interventions: Combination Product: Transarterial chemoembolization
- Arm 3 - DEB - CLOSED (Experimental): Lobar or segmental hepatic chemoembolization with DEBDOX (100-300 or 300-500 micron beads loaded with doxorubicin per manufacturer IFU monthly until entire tumor burden is treated.
  Interventions: Combination Product: Drug Eluting Beads Embolization

INTERVENTIONS:
Device: Bland Embolization — Lobar or segmental bland embolization with microspheres (50-500 microns) to 2-5 heartbeat stasis
  Other Names: BE
  Arms: Arm 1 - BE
Combination Product: Transarterial chemoembolization — Lobar or segmental lipiodol transarterial chemoembolization. Doxorubicin 50 mg dissolved in 10 mL dilute contrast and emulsified with 10-20 cc iodized oil, followed by 50-500 μm microspheres.
  Other Names: TACE
  Arms: Arm 2 - TACE
Combination Product: Drug Eluting Beads Embolization — CLOSED - Lobar or segmental hepatic chemoembolization with DEBDOX (100-300 or 300-500 micron beads loaded with doxorubicin per manufacturer IFU.
  Other Names: DEB
  Arms: Arm 3 - DEB - CLOSED

SUMMARY:
The primary aim of this trial is to estimate the duration of hepatic progression-free survival (HPFS) in participants treated with bland embolization (BE), transcatheter arterial Lipiodol chemoembolization (TACE), and embolization by drug-eluting beads (DEB). The primary hypothesis is that chemoembolization will be nearly twice as durable as bland embolization; thatis, the hazard ratio for HPFS will be 1.76 or better.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 years and older;
* Biopsy-proven neuroendocrine tumor.
* Measurable metastasis to liver with at least one dimension ≥ 1.0 cm.
* Tumor burden dominant in the liver AND liver tumor burden less than or equal to 70% of the total liver volume by visual estimate.
* Not a candidate for surgical resection based on unresectability, anatomy, anesthesia risk, patient preference.
* Symptoms uncontrolled by somatostatin analogues OR morphologically progressive tumor by RECIST 1.1 criteria in the liver OR baseline tumor burden >25% of the liver volume.
* There must be no plans for the patient to receive other concomitant therapy while on this protocol treatment (other than somatostatin analogs or bone-strengthening agents).
* Performance status 0-2 on Zubrod/ECOG Performance Scale;
* Serum creatinine < 2.0 mg/dL;
* Serum Bilirubin ≤ 2.0 mg/dL
* Serum albumin ≥ 3.0 g/dL
* Platelet count > 50 thousands/uL (corrected if needed)
* INR ≤ 1.5 (corrected if needed)
* All patients must be informed of the investigational nature of this study and must sign a study specific informed consent in accordance with institutional and federal guidelines prior to study entry.

Exclusion Criteria:

* Pregnant or lactating women may not participate due to the embryotoxic effects of protocol treatment. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Prior hepatic arterial therapy or hepatic radiation therapy. Prior surgical resection or ablation of liver metastases is acceptable. Patients must be at least one month beyond prior chemotherapy, PRRT, ablation or surgery, and have recovered from all therapy-associated toxicities.
* Active infection (Symptomatic bacterial and fungal infection - newly diagnosed and/or requiring treatment);
* Choledochoenteric anastomosis; transpapillary biliary stent, or sphincterotomy of duodenal papilla
* Absolute contraindication to intravenous iodinated contrast (Hx of significant previous contrast reaction, not mitigated by appropriate pre-medication).
* Contraindications to arteriography and selective visceral catheterization:

  1. severe allergy or intolerance to contrast media, narcotics, sedatives, or atropine.
  2. bleeding diathesis not correctable by usual forms of therapy.
  3. severe peripheral vascular disease precluding catheterization.
* Contraindications to hepatic artery embolization:

  1. portal vein occlusion without hepatopedal collateral flow demonstrated by angiography; or portal hypertension with hepatofugal flow.
  2. hepatic encephalopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Abdominal MRI/Triple Phase CT | 2 years
  Hepatic progression-free interval (H-PFS)

SECONDARY OUTCOMES:
Number of Adverse Events | 2 years
  Symptom-relief interval and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Soulen, MD, FSIR, Principal Investigator — University of Pennsylvania
Locations (13):
- United States (10):
  - University of California San Francisco, San Francisco, California
  - Stanford University, Standford, California
  - Moffitt Cancer Center, Tampa, Florida
  - Mount Sinai School of Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen JX, Wileyto EP, Soulen MC. Randomized Embolization Trial for NeuroEndocrine Tumor Metastases to the Liver (RETNET): study protocol for a randomized controlled trial. Trials. 2018 Jul 17;19(1):390. doi: 10.1186/s13063-018-2782-5. PMID 30016989